CLINICAL TRIAL: NCT05554939
Title: A Phase 1/2 Clinical Trial of Gene-edited Allogenic CD19 Targeting Chimeric Antigen Receptor-γδT Cells Therapy in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Allogenic CD19-targeting CAR-γδT Cell Therapy in R/R NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-072
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Non Hodgkin's Lymphoma
Keywords: B-cell malignancies; Relapsed or refractory; CD19 CAR-γδT
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory or relapsed B-cell NHL (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, allogenic targeting CD19 chimeric antigen receptor γδT cells.
  Interventions: Biological: Allogenic CD19 CAR-γδT cell; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Allogenic CD19 CAR-γδT cell — Phase 1 dose escalation (3+3) : dose 1 (6 × 10^6 cells/kg) , dose 2 (1.2 × 10^7 cells/kg), dose 3 (1.8 × 10^7 cells/kg); Phase 2 : dose of RP2D.
Drug: Fludarabine — Intravenous fludarabine 30~50 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 500~1000 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
This is a single center, prospective, open-label, single-arm, phase 1/2 study for patients with r/r B-cell NHL to evaluate the safety and efficacy of gene edited allogenic CD19 CAR-γδT cells. The cells are from healthy adult volunteer donors that are gene edited ex vivo using CRISPR-Cas9 to weaken HLA expression and further to overcome host immune system rejection (HvGR). In this study, a second generation anti-CD19 CAR prototype was constructed, bearing murine FMC63 single-chain variant fragment (scFv) together with intracellular 4-1BB co-stimulatory and CD3ζ signaling domains linked by a CD8α sequence comprising the hinge and transmembrane domains.

A total of around 30 patients with r/r B-cell NHL will be enrolled in the study and receive allogeneic CD19 CAR-γδT cell infusion. Phase 1 (n=9 to 12) is dose escalation part, and phase 2 (n=15 to 20) is expansion cohort part. The primary objective of this study was to evaluate the safety and efficacy of allogeneic CD19 CAR-γδT cell therapy in patients with r/r B-cell NHL.

DETAILED DESCRIPTION:
Phase 1 (dose escalation)

In phase 1, 9-12 subjects will be enrolled. Subjects will receive 3 doses of CD19 CAR- γδ T cell therapy (6 × 10^6 cells/kg、1.2× 10^7 cells/kg、1.8 × 10^7 cells/kg) increases from low dose to high dose according to the "3 + 3" principle:

1. Three patients were enrolled in the lowest dose group.
2. Subsequent patients were enrolled according to the following rules:

   1. If the incidence of dose limiting toxicity (DLT) was 0/3, 3 patients were enrolled in the next high-dose group.
   2. If the incidence of DLT was 1/3, 3 patients were enrolled at the same dose; If the incidence of DLT was 1/3 + 0/3, 3 patients were enrolled in the next high-dose group. If the incidence of DLT was 1/3 + 1/3, this dose was defined as maximum tolerated dose (MTD); If the incidence of DLT was 1/3 + 2/3 or 1/3 + 3/3, the previous dose was MTD.
   3. If the incidence of DLT was 2/3 or 3/3, the previous dose was MTD.

To ensure the safety of the subjects, the first subject in each dose group was observed for at least 28 days after the cell infusion. If no DLT occurred, the remaining two subjects could be enrolled and treated at the same dose level. The safety data of all subjects in each dose group until day 28 should be reviewed and tolerated before proceeding to the next dose group trial. No dose escalation was allowed for the same subject during the trial. If a subject drop out during the observation period due to non-DLT reasons, new subjects should be enrolled to make up for the number of subjects who drop out.

Phase 2 (expansion cohort)

In phase 2, 15 to 20 subjects will be enrolled and receive CD19 CAR-γδ T cell infusion at dose of RP2D, which will be determined based on the MTD, occurrence of DLT, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.

Objectives

The primary objectives of the phase 1 were to evaluate the tolerability, safety, and determine recommended phase 2 dose (RP2D). The primary purpose of the phase 2 study was to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria for patients:

1. Age 18-75 (inclusive).
2. Patients with histologically confirmed CD19-positive B-cell NHL, including the following types defined by the World Health Organization (WHO) 2016:

   * Diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS), including Activated B-cell type (ABC）/Germinal center B-cell type（GCB）;
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
   * Transformed follicular lymphoma (TFL);
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
   * Follicular lymphoma (FL);
   * Mantle cell lymphoma (MCL) (pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1);
   * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.
3. Relapse after treatment with ≥2 lines systemic therapy for all the above disease types, or refractory disease for aggressive types (DLBCL-NOS, PMBCL, TFL and HGBCL). Relapse disease is defined as disease progression after last regimen. Refractory disease is defined as no CR to first-line therapy:

   * PD as best response to first-line therapy, or
   * SD as best response after at least 4 cycles of first-line therapy (eg,4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT) i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.
4. Individuals must have received adequate prior therapy:

   * For MCL, prior therapy must have included:

     * Anthracycline or bendamustine-containing chemotherapy and
     * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
     * Bruton's tyrosine kinase inhibitor (BTKi)
   * For other types, prior therapy must have included:

     * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
     * Anthracycline containing chemotherapy regimen.
   * For individual with transformed FL must have relapse or refractory disease after transformation to DLBCL.
5. The estimated survival time is over 3 months.
6. The Eastern Cooperative Oncology Group (ECOG) score is 0-2.
7. According to Lugano response criteria 2014, there should be at least one evaluable tumor focus. Evaluable tumor focus was defined as that with the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
8. Subjects must be willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
9. Functions of important organs meet the following requirements: Echocardiography showed left ventricular ejection fraction ≥50%. Serum creatinine ≤1.5 × upper limit of normal range (ULN) or endogenous creatinine clearance ≥45mL/min (cockcroft-gault formula); Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤3 times ULN, Total bilirubin ≤1.5× ULN; Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
10. Blood routine (normal values shall not be obtained with growth factors, and hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions below): hemoglobin (Hgb) ≥80g/L, neutrophil count≥1×10^9/L, platelet (PLT) ≥75×10^9/L.
11. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
12. Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
13. No obvious hereditary diseases.
14. Able to understand the requirements and matters of the trial, and willing to participate in clinical research as required.
15. Informed consent must be signed.

Exclusion Criteria for patients:

1. During the screening period, there was central nervous system (CNS) invasion or a history of clinically significant central nervous system diseases, such as epilepsy and cerebrovascular diseases.
2. Women who are pregnant or breastfeeding, or who do not agree to use effective contraception during treatment and during the subsequent 1 year.
3. History of allogeneic hematopoietic stem cell transplantation, or organ transplantation.
4. History of other malignancies that have not been in remission.
5. Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy.
6. Received radiotherapy within 3 months before enrollment.
7. Received immunotherapy drugs within 4 weeks before enrollment, such as anti-programmed death 1 (PD-1) antibody, anti-programmed death ligand 1 (PD-L1) antibody, CD19/CD3-bispecific antibody, and so on.
8. Patients who received any immunocellular therapy within 3 months before enrollment.
9. Confirmed evidence showing positiveness of anti-CD19 scFv reaction in patient serum.
10. Patients who participated in other clinical trials within 4 weeks prior to enrollment.
11. Uncontrolled infectious diseases or other serious illnesses, including but not limited to infections [e.g., human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B (HBV) or C (HCV) infection], congestive heart failure, unstable angina, arrhythmias, or that pose an unpredictable risk in the opinion of the attending physician.
12. The presence of uncontrollable serous membrane fluid, such as massive pleural effusion or ascites.
13. A history of stroke or intracranial hemorrhage within 3 months prior to enrollment.
14. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
15. Received allogeneic cell therapy within 6 weeks prior to enrollment, such as donor lymphocyte infusion.
16. History of allergies to any of the ingredients in cell products.
17. Conditions in which a known mental or physical illness interferes with cooperation with the requirements of the study or disrupts the results or interpretation of the results and, in the opinion of the therapeutic investigator, makes the patient unfit for study participation.
18. There is the situation that the researcher's judgment will interfere with the whole study participation; Situations where there is significant risk to the subject; Or interferes with the interpretation of research data.
19. Inability to understand or unwillingness to sign informed consent.
20. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of lymphodepletion to 12 months after CD19 CAR-γδT cells infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versus-host disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1: Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of CD19 CAR-γδT cells up to 28 days
  DLT was defined as CD19 CAR-γδT cells-related events with onset within first 28 days following infusion:
  * Grade 3 aGVHD that does not resolve to Grade 1 or 2 within 7 days, with the exception of isolated skin involvement aGVHD;
  * Grade 4 CRS or grade 3 CRS that does not resolve to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥7 days or Grade 4 ICANS;
  * Any other Grade ≥4 and Grade 3 AE related to the CAR-γδT that lasts for ≥14 days, except hematology toxicity.
Phase 1: Recommended Phase 2 Dose (RP2D) | 12 months
  The recommended dose for phase 2 was determined through phase 1 study.
Phase 2: Best Objective Response Rate | 24 months
  The incidence of complete response (CR) and partial response (PR) as the best response to treatment assessed by investigatorand based on the Lugano 2014 assessment criterion.
Phase 2: Best Complete Response Rate | 24 months
  The incidence of complete response (CR) as the best response to treatment assessed by investigatorand based on the Lugano 2014 assessment criterion.

SECONDARY OUTCOMES:
Phase 2: Overall Survival (OS) | 24 months after the first infusion of CD19 CAR-γδT cells
  OS is defined as the time from CD19 CAR-γδT cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months after the first infusion of CD19 CAR-γδT cells
  PFS is defined as the time from the CD19 CAR-γδT cells infusion to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Phase 2: Time to Response (TTR) | 24 months
  TTR is defined as the time from CD19 CAR-γδT infusion to first assessed CR or PR by investigators and based on the Lugano 2014 assessment criterion.
Phase 2: Duration of Response (DOR) | 24 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B-cell NHL, or death regardless of cause.
Pharmacokinetics: Number and Copy Number of CD19 CAR-γδT cells (phase 1 and phase 2) | 12 months
  Number and copy number of CD19 CAR-γδT cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CD19 CAR-γδT cells were not detected for two consecutive times) to detect the number and copy number of CD19 CAR-γδT cells, and to evaluate the pharmacokinetics of CD19 CAR-γδT.
Pharmacokinetics: Persistence of CD19 CAR-γδT (phase 1 and phase 2) | 12 months
  Persistence of CD19 CAR-γδT cell assessed by number in peripheral blood.
Pharmacodynamics: Peak Level of Cytokines in Serum (phase 1 and phase 2) | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.

OTHER OUTCOMES:
Correlation Between Infusion Dose of CD19 CAR-γδT Cells and Efficacy | 12 months
  Efficacy was assessed using the objective response rate. The correlation between infusion dose and efficacy was analyzed by calculating the ORR in different dose groups.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (2):
- China (2):
  - School of phamaceutical, Tsinghua University, Beijing, Beijing Municipality
  - Biotherapeutic Department, Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No